CLINICAL TRIAL: NCT00410774
Title: A Phase I/II Study of Fixed-Dose Rate Gemcitabine and Bevacizumab for Postoperative Adjuvant Treatment of Patients With Resected Pancreatic Cancer
Brief Title: Gemcitabine and Bevacizumab in Treating Patients With Pancreatic Cancer That Has Been Completely Removed By Surgery
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low accrual-no data available
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000517330; UCSF-06451; UCSF-H12191-28980-01
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; stage I pancreatic cancer; adenocarcinoma of the pancreas; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Gemcitabine; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: bevacizumab
Drug: gemcitabine hydrochloride
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of pancreatic cancer by blocking blood flow to the tumor. Giving gemcitabine and bevacizumab after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase I/II trial is studying the side effects of gemcitabine and bevacizumab and to see how well they work in treating patients with pancreatic cancer that has been completely removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of adjuvant, fixed-dose rate gemcitabine hydrochloride and bevacizumab in patients with completely resected pancreatic cancer.
* Determine the 1-year disease-free survival rate in patients treated with this regimen.

Secondary

* Determine the 1- and 2-year overall survival rates in these patients.
* Determine the median disease-free survival rate in these patients.
* Determine the median overall survival rate in these patients.

OUTLINE: This is an open-label, non-randomized study.

Patients receive gemcitabine hydrochloride IV over 100 minutes followed by bevacizumab* IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease recurrence or unacceptable toxicity.

NOTE: *The first dose of bevacizumab is not administered until after 6 weeks have passed since surgery.

After completion of study therapy, patients are followed periodically for 18 months.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Completely resected disease

    * Underwent 1 of the following procedures 3-8 weeks ago:

      * Standard pancreaticoduodenectomy (for tumors of the pancreatic head)
      * Distal pancreatectomy (for tumors of the pancreatic tail)
    * No grossly positive surgical margins

      * Positive microscopic margins allowed
* Nonmeasurable disease
* No known CNS disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy
* CA 19-9 ≤ 2.5 times upper limit of normal (ULN)
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin ≥ 9 g/dL (transfusion or epoetin alfa allowed)
* Platelet count ≥ 100,000/mm³
* INR ≤ 1.5 (except in patients receiving full-dose warfarin)
* Bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 2.0 mg/dL
* No clinically significant impairment of renal function
* No postoperative complications, including any of the following:

  * Wound dehiscence or infection
  * Intra-abdominal abscess
  * Pancreatic or biliary leak or fistula
  * Grade 3 or 4 delayed hemorrhage (occurring > 5 days postoperatively)
  * Bowel perforation
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abcess within the past 6 months
* No history of major psychiatric disorder or other chronic medical illness that, in the opinion of the treating physician, contraindicates use of the study drugs or renders the patient at high risk of treatment-related complications
* No other cancer within the past 5 years except basal cell or squamous cell skin cancer
* No history of serious systemic disease, including any of the following:

  * Myocardial infarction or unstable angina within the past 12 months
  * New York Heart Association class II-IV congestive heart failure
  * Unstable symptomatic arrhythmia requiring medication

    * Chronic atrial arrhythmia (i.e., atrial fibrillation or paroxysmal supraventricular tachycardia) allowed
* No history of stroke or transient ischemic attack
* No symptomatic peripheral vascular disease
* No significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* No inadequately controlled hypertension (i.e., blood pressure > 150/100 mm Hg on antihypertensive medication)
* No prior hypertensive crisis or hypertensive encephalopathy
* No proteinuria (defined as urine protein:creatinine ratio ≥ 1.0 OR proteinuria ≥ 2+ by dipstick urinalysis OR protein > 1 g by 24-hour urine collection)
* No serious, nonhealing wound or ulcer
* No evidence of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 28 days

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or radiotherapy for pancreatic cancer
* No prior systemic or investigational therapy for pancreatic cancer
* No major surgical procedure (except for resection of pancreatic cancer) or open biopsy within the past 28 days
* No fine-needle aspiration or core biopsy within the past 7 days
* No anticipated need for a major surgical procedure during study treatment
* No concurrent newly prescribed nonsteroidal anti-inflammatory drugs (NSAIDs)

  * Concurrent chronic-dose NSAIDs for analgesia are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety of gemcitabine when administered with bevacizumab as assessed by NCI CTCAE v3.0
Disease-free survival rate at 1 year

SECONDARY OUTCOMES:
Overall survival rate at 1 and 2 years
Median disease-free survival rate at 1 and 2 years
Median overall survival rate at 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ko, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States